CLINICAL TRIAL: NCT05509231
Title: Effects of a Multimodal Exercise Program for Children With Autistic Spectrum Disorder (ASD) on Cognitive and Motor Abilities: Part III
Brief Title: Effects of a Multimodal Exercise Program for Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1599
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder; Asperger Syndrome
Keywords: Developmental Coordination Disorder; Dyspraxia; Dysgraphia; Incoordination; Motor control
MeSH Terms: conditions — Autism Spectrum Disorder; Asperger Syndrome; Motor Skills Disorders; Apraxias; Agraphia; Ataxia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will consist of individuals diagnosed with autism spectrum disorder and neurotypical children. The intervention includes high-intensity whole-body exercise (Group 1), intervention using wearable technology (arm and sleeve sensor) (Group 2), and no-intervention control (waitlist control) (Group 3). Experienmental Group 1 will participate in a traditional physical fitness program combined with exergaming, Group 2 will train using wearable technology, and Group 3 will be waitlisted for the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ASD High-intensity Exercise (Group 1a - ASD) (Experimental): The high-intensity group (Group 1a - ASD). Subjects will be asked to meet 2-3 times a week for exercise training for 60-90 minutes a session. Subjects will be asked to take part in tests that measure motor skills and thinking abilities.
  Interventions: Behavioral: High-intensity exercise
- Neurotypical Group (Group 1b - Neurotpical) (Experimental): The high-intensity group (Group 1b - Neurotypical). Subjects will be asked to meet 2-3 times a week for exercise training for 60-90 minutes a session. Subjects will be asked to take part in tests that measure motor skills and thinking abilities.
  Interventions: Behavioral: High-intensity exercise
- ASD Wearable Technology (Group 2a - ASD) (Experimental): ASD Wearable Technology (Group 2a- ASD). Subjects wear a glove and arm sleeve with sensors that will measure arm and hand performance. Subjects will be training 2 times a week for 20-30 minutes. The Subjects will be asked to copy a series of hand and arm gestures. Subjects will perform a series of hand exercises with the glove. The glove will record the movement data that will provide the investigators and subjects feedback on hand performance and fine motor capabilities.
  Interventions: Device: Wearable glove and arm sleeve device to measure movement
- ASD Wearable Technology (Group 2b - Neurotypical) (Experimental): ASD Wearable Technology (Group 2b - Neurotypical). Subjects wear a glove and arm sleeve with sensors that will measure arm and hand performance. Subjects will be training 2 times a week for 20-30 minutes. The Subjects will be asked to copy a series of hand and arm gestures. Subjects will perform a series of hand exercises with the glove. The glove will record the movement data that will provide the investigators and subjects feedback on hand performance and fine motor capabilities.
  Interventions: Device: Wearable glove and arm sleeve device to measure movement
- Control (Group 3) (No Intervention): The wait-list control group will not receive the experimental intervention but will be put on a waiting list to receive the intervention after the active intervention group completes the study.

INTERVENTIONS:
Behavioral: High-intensity exercise — Gross motor physical fitness activities to improve proprioceptive awareness, motor control, and coordination.
  Other Names: Gross motor physical fitness
  Arms: ASD High-intensity Exercise (Group 1a - ASD); Neurotypical Group (Group 1b - Neurotpical)
Device: Wearable glove and arm sleeve device to measure movement — Sign language and other fine motor skills activities using wearable technology.
  Arms: ASD Wearable Technology (Group 2a - ASD); ASD Wearable Technology (Group 2b - Neurotypical)

SUMMARY:
Exploring the effects of an exercise program for children ages 6 -26 years old who have been diagnosed with autism spectrum disorder and neurotypical children respond to high-intensity whole body exercise interventions (Group 1), training using a sensory glove and armband (Group 2), no-intervention control (waitlist control) (Group 3). Approximately 50 children and adolescents will volunteer to participate in this program with participants parents' (or legal guardians') permission. This study will be conducted at an off-site pediatric occupational therapy facility Inclusive Sports and Fitness, Inc. (ISF).

DETAILED DESCRIPTION:
The purpose of this study is to explore the effects of a structured high-intensity sensorimotor exercise program on performance skills (cognitive or executive function and functional motor skills) and hand function of children diagnosed with autistic spectrum disorder (ASD) and a neurotypical group and an additional qEEG which will be administered during the 6-12 week period. The investigators would like to recruit 50 participants for this study.

The research design consists of a nonequivalent quasi-experimental multi-group (ASD and Neurotypical) pre and post-test group design: Experimental Group 1 (high-intensity whole-body exercise): Pretest - intervention - Post-test; Experimental Group 2 (Sensory glove and armband): Pretest-Intervention-Post-test. The pretest will consist of motor and cognitive testing and a quantitative electroencephalogram (qEEG). The administration of these measures will be conducted on the grounds of the clinical site (ISF). The same measures used at the pretest will be utilized during post-test.

The potential benefits from the findings of this study will provide important information as to the efficacy of using multimodal (multisensory) training with exergaming applications on performance skills and abilities. The multisensory feedback will come from a number of sensory-based activities and gaming mechanisms employed in occupational and physical therapy. To our knowledge, there is a limited number of studies in peer-reviewed literature using validated and reliable outcome assessments under scientifically rigorous methods. The children participating in this study will receive the benefits of being in a skill-oriented exercise and functional skills training program that will address their performance skills impairments. These types of programs are not available to this population, particularly for families with limited financial support. Cognitive interventions will address the participants' ability to process various sensory (visual, auditory, haptic, proprioceptive, and vestibular information. The intervention will include a combination of cognitive tasks and sensorimotor activities. The investigators are utilizing a dynamic system approach that integrates sensory, physical, and cognitive processes with wearable technology and gaming. This approach recognizes the plastic nature of the brain and its ability to adapt through skilled interventions. Recent studies have posited that the neural substructures associated with functional impairments in children with ASD are not localized to morphological brain disorders, but rather a connectome issue associated with interneuron network impairments. Disordered connectivity can impair information processing, integration, and application of information from the different "processing nodes" within a functional network. Children with ASD demonstrate poor integration of multisensory information utilizing qEEG. The researchers suggested that interventions that provide multisensory stimuli may help improve neural connections and help them develop strategies for functioning in mainstream environments. In addition to the multisensory interventions to advance interconnectivity in the brain, children will participate in high-intensity physical activity. High-intensity activity has been found to produce neurophysiological and morphological changes in the brain with subsequent cognitive improvements.

Test and measures will be administered using the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2). The BOT-2 covers the age range of 4 to 21 years, with a 53-item assessment consisting of eight subtests designed as game-like tasks that measure hand and arm coordination, balance, mobility, and strength. Investigators will be including an assessment that will allow us to measure the quality of movement of the hand. It will also provide feedback to the user to better calibrate and isolate hand movements. The participant will don a glove and arm sleeve with inductive sensors that will measure hand performance. The participants are asked to make a series of hand gestures for numbers 1 to 9 based on the American Sign Language and then follow some patterns of arm movements. The glove will record the kinematic data corresponding to each hand gesture and arm movement using a set of inductive sensors in the form of patches to be attached to the arm, a glove, and/or a pad of inductive sensors. The data will be used to develop machine learning algorithms from the gestures and arm movements made by neurotypical and ASD children and young adults. Machine learning applications will provide user feedback to identify correct hand positions and improve fine motor capabilities.

Cognitive Performance Measure The Test of Variables of Attention (TOVA). The TOVA is a culture- and language-free, sufficiently long computerized test that requires no left/right discrimination or sequencing. Responses to visual or auditory stimuli are recorded with a unique, highly accurate (±1 ms) microswitch. The TOVA calculates response time variability (consistency), the response time (speed), commissions (impulsivity), and omissions (focus and vigilance). These calculations are then compared to a large age- and gender-matched normative sample, as well as to a sample population of individuals independently diagnosed with ADHD.

Qualitative EEG (qEEG) Those potential participants who meet the eligibility criteria of the screening visit will be invited to participate in the study. As a baseline, qEEG will be a measure and guide in the individualized intervention protocol group. The qEEG is used to study a person's brainwaves via an analytic procedure called "brain mapping." The qEEG is derived by digitally analyzing the EEG to measure the amount of various EEG frequencies at different scalp locations (power analysis) and the connections between different areas (coherence analysis). Quantitative EEG frequencies will be measured at 19 sites on the head. The data obtained at 19 standard sites on the head is compared with data from normal individuals in the Applied Neuroscience, Inc. database. qEEG data will be analyzed to obtain brain maps and Z Scores for each participant. These qEEG analyses will provide a baseline for before/during/after intervention comparison in the individualized intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Autism Spectrum Disorder (ASD)

   * Level 1 or Level 2
2. Neuro-typical individual with no history of developmental disabilities
3. Medical clearance to participate in the physical fitness activities

Exclusion Criteria:

1. Diagnosis of Autism Spectrum Disorder (ASD)

   * Level 3
2. Nonverbal
3. IQ below 80 as assessed by the Wechsler Abbreviated Scale of Intelligence
4. History of seizures or head trauma; and any medical condition that precludes participants from participating in physical fitness activities.

Ages: 6 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-12 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) | 60 minutes
  Bruininks-Oseretsky Test of Motor Proficiency (BOT-2). The BOT-2 covers the age range of 4 to 21 years, with a 53-item assessment consisting of eight subtests designed as game-like tasks that measure hand and arm coordination, balance, mobility, and strength.

SECONDARY OUTCOMES:
Qualitative EEG (qEEG) | 10 minutes
  As a baseline, qEEG will be a measure and guide in the individualized intervention protocol group. The qEEG is used to study a person's brainwaves via an analytic procedure called "brain mapping." The qEEG is derived by digitally analyzing the EEG to measure the amount of various EEG frequencies at different scalp locations (power analysis) and the connections between different areas (coherence analysis). Quantitative EEG frequencies will be measured at 19 sites on the head. The data obtained at 19 standard sites on the head is compared with data from normal individuals in the Applied Neuroscience, Inc. database. qEEG data will be analyzed to obtain brain maps and Z scores for each participant. These qEEG analyses will provide a baseline for before/during/after intervention comparison in the individualized intervention group. Furthermore, data obtained through qEEG before and after interventions will be used to evaluate the progress and modulation of brain functional connectivity.
Wearable technology: Glove and armband | Approximately 20-30 minutes
  The assessment requires the donning of a glove and armband with inductive sensors that will measure hand performance. The participants are asked to make a series of hand gestures for numbers 1 to 9 based on the American Sign Language and then follow some patterns of arm movements. The glove will record the kinematic data corresponding to each hand gesture and arm movement using a set of inductive sensors in the form of patches to be attached to the arm, a glove, and/or a pad of inductive sensors.

OTHER OUTCOMES:
Kinematic Assessment with Glove and Arm Band | Approximately 10-20 minutes
  We will be including an assessment that will allow us to measure the quality of movement of the hand. It will also provide feedback to the user to better calibrate and isolate hand movements. The subjects will don a glove and arm sleeve with inductive sensors that will measure hand performance. The subjects are asked to make a series of hand gestures for numbers 1 to 9 based on the American Sign Language and then follow some patterns of arm movements. The glove will record the kinematic data corresponding to each hand gesture and arm movement using a set of inductive sensors in the form of patches to be attached to the arm, a glove, and/or a pad of inductive sensors. The data will be used to develop machine learning algorithms from the gestures and arm movements made by neurotypical and ASD children and young adults. Machine learning applications will provide user feedback to identify correct hand positions and improve fine motor capabilities.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] David FJ, Baranek GT, Giuliani CA, Mercer VS, Poe MD, Thorpe DE. A pilot study: coordination of precision grip in children and adolescents with high functioning autism. Pediatr Phys Ther. 2009 Summer;21(2):205-11. doi: 10.1097/PEP.0b013e3181a3afc2. PMID 19440131
- [Background] Brandwein AB, Foxe JJ, Butler JS, Russo NN, Altschuler TS, Gomes H, Molholm S. The development of multisensory integration in high-functioning autism: high-density electrical mapping and psychophysical measures reveal impairments in the processing of audiovisual inputs. Cereb Cortex. 2013 Jun;23(6):1329-41. doi: 10.1093/cercor/bhs109. Epub 2012 May 24. PMID 22628458
- [Background] Hillman CH, Snook EM, Jerome GJ. Acute cardiovascular exercise and executive control function. Int J Psychophysiol. 2003 Jun;48(3):307-14. doi: 10.1016/s0167-8760(03)00080-1. PMID 12798990
- [Background] Rogers RL, Meyer JS, Mortel KF. After reaching retirement age physical activity sustains cerebral perfusion and cognition. J Am Geriatr Soc. 1990 Feb;38(2):123-8. doi: 10.1111/j.1532-5415.1990.tb03472.x. PMID 2299115
- [Result] Baio J, Wiggins L, Christensen DL, Maenner MJ, Daniels J, Warren Z, Kurzius-Spencer M, Zahorodny W, Robinson Rosenberg C, White T, Durkin MS, Imm P, Nikolaou L, Yeargin-Allsopp M, Lee LC, Harrington R, Lopez M, Fitzgerald RT, Hewitt A, Pettygrove S, Constantino JN, Vehorn A, Shenouda J, Hall-Lande J, Van Naarden Braun K, Dowling NF. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2014. MMWR Surveill Summ. 2018 Apr 27;67(6):1-23. doi: 10.15585/mmwr.ss6706a1. PMID 29701730
- [Result] Liu H, Song L, Zhang T. Changes in brain activation in stroke patients after mental practice and physical exercise: a functional MRI study. Neural Regen Res. 2014 Aug 1;9(15):1474-84. doi: 10.4103/1673-5374.139465. PMID 25317160
- [Result] Arslan E, Ince G, Akyuz M. Effects of a 12-week structured circuit exercise program on physical fitness levels of children with autism spectrum condition and typically developing children. Int J Dev Disabil. 2020 Sep 17;68(4):500-510. doi: 10.1080/20473869.2020.1819943. eCollection 2022. PMID 35937176
- [Result] Fuentes CT, Mostofsky SH, Bastian AJ. Children with autism show specific handwriting impairments. Neurology. 2009 Nov 10;73(19):1532-7. doi: 10.1212/WNL.0b013e3181c0d48c. PMID 19901244
- [Result] Mostofsky SH, Ewen JB. Altered connectivity and action model formation in autism is autism. Neuroscientist. 2011 Aug;17(4):437-48. doi: 10.1177/1073858410392381. Epub 2011 Apr 5. PMID 21467306
- [Result] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2008 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--Autism and Developmental Disabilities Monitoring Network, 14 sites, United States, 2008. MMWR Surveill Summ. 2012 Mar 30;61(3):1-19. PMID 22456193
- [Result] Muller RA. The study of autism as a distributed disorder. Ment Retard Dev Disabil Res Rev. 2007;13(1):85-95. doi: 10.1002/mrdd.20141. PMID 17326118
- [Result] Yanagisawa H, Dan I, Tsuzuki D, Kato M, Okamoto M, Kyutoku Y, Soya H. Acute moderate exercise elicits increased dorsolateral prefrontal activation and improves cognitive performance with Stroop test. Neuroimage. 2010 May 1;50(4):1702-10. doi: 10.1016/j.neuroimage.2009.12.023. Epub 2009 Dec 16. PMID 20006719